CLINICAL TRIAL: NCT05218993
Title: A New Dual Task Capacity Measuring Method for Football Players
Brief Title: A New Dual Task Test Method for Football Players
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgün Uysal, Principal Investigator, Hacettepe University
Other Study IDs: DualTask
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Sports Physical Therapy; Multi-Tasking Behavior; ACL Injury; Kinesiophobia
Keywords: soccer; dual task; performance; rehabilitation; return to sport
MeSH Terms: conditions — Multitasking Behavior; Anterior Cruciate Ligament Injuries; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Development of the new dual task test: the new two different method of dual task measurement and a traditional dual task measurement method and also, cognitive and performance measurement test will be conducted.
  Interventions: Diagnostic Test: A new dual-task measurement method with images; Diagnostic Test: A new dual-task measurement method with cards
- Collecting the normative values: Better dual task measurement method (from the two methods) will be conducted at different football levels.
  Interventions: Diagnostic Test: A new dual-task measurement method with images; Diagnostic Test: A new dual-task measurement method with cards
- Measurement of the athletes in return to sport stage: new dual task measurement method and other return to sport measurements will be conducted on athletes who wish to return to sport.
  Interventions: Diagnostic Test: A new dual-task measurement method with images; Diagnostic Test: A new dual-task measurement method with cards

INTERVENTIONS:
Diagnostic Test: A new dual-task measurement method with images — Football players will perform Illinois t test with and without cognitive demand with images. These images will represent scenarios from football with some of the players in the scene are from his team and others from opposing team. The player will be asked to look at the image and say the number on the player in following scenarios; The player to whom he can pass the ball, The player who is most likely to intervene the ball, The player who can score the goal. In order to reduce the other possibilities, opposing team players will be positioned in a specific way to block all team-mates but one.
Diagnostic Test: A new dual-task measurement method with cards — Football players will perform Illinois t test with and without cognitive demand with cards and balls. On the path of Illinois t test, there will be 3 football balls, 3-meters apart from each other, and there will be cards behind each, which can only be seen when the player about to hit the ball. This cards will vary in color (blue or red), which mean right or left. If the player sees red card, he will shoot the ball to the left side goal and if the player sees blue card, he will shoot the ball to the right side.

SUMMARY:
Multitasking (Dual Task) is a measurement method to evaluate cognitive ability to execute multiple functions at the same time. To perform this test, while participant/patient performing a main skill (for example, walking), a cognitive skill is added (for example, counting 7 backwards from 100) to measure how much the completion performance of the activity is affected. Frequently used multitasking trainings are known as counting back from 100 and asking mathematical equations during a physical skill. Multitasking skill is rarely used in sports-related training, and it is generally used in the form of counting 7 backwards from 100, counting months and counting 5-letter words while walking over obstacles. However, multitasking training methods described and applied in the literature are not specific to football skills. For this reason, limited tests defined and applied in other clinical and sportive fields may not be sufficient in football players who perform activities that require high performance. Therefore, aim of this study is to develop a dual-task assessment method, which includes the cognitive loads experienced by football players during training and matches, and also covers the basic skills of football. As a result of this study, a football-specific dual-task test will be created and the capacity of the athletes will be measured by applying this test to healthy athletes. Also, this test will be conducted on football players with recent knee injury history, who wish to return to sport, and to evaluate their dual-task capacity and to correlate it with kinesiophobia and other performance tests

ELIGIBILITY:
Inclusion Criteria:

* attending regularly to the trainings
* being a professional football player

Exclusion Criteria:

* having any neurological disorders

Min Age: 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For the first stage of the study, professional football players who are healthy and who can attend the trainings and/or games in full performance.
  For the last stage of the study, professional football players who wish to return to sports after knee injuries.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Traditional dual task assessment | At the baseline
  Players will dribble with the ball with and without cognitive task. As cognitive task, players would be asked to count down from 100, by 7.

SECONDARY OUTCOMES:
Juggling tests | At the baseline
  Player will juggle the ball with both feet as much as he can, until the count of 25. Best of right and left foot will be recorded. For the second trial, player will juggle the ball in all of the following orders: chest-foot-head, head-left foot-right foot or foot-chest-head. Each correct trial scores as 1 point and total of 9 points can be taken.
Fast dribbling test | At the baseline
  Player would dribble through an obstacle course as much as they can and the total time is recorded.
Long pass accuracy test | At the baseline
  Player will be asked to long pass the ball in to a 2m-radius circle within a 10m by 10m square from 36 meters distance. 3 points is scored if ball falls within the circle and 1 points is scored if the ball falls within the square. Total of 5 repetitions is recorded.
Stroop test | At the baseline
  There will be color names appearing on the computer screen written in different color (for example: word "yellow" written in blue) and player is asked to pick the name of the color. total time to correctly pick 10 names is measured and recorded.
Corsi task | At the baseline
  From the 9 balls appearing on the screen, three of them will blink in random order. Player will be asked to click on them in the same order of blinking. For each correct trial, the number of blinking balls will increase until all of the balls are blinking. total number of right order will be recorded.
Simple and choice based reaction times | At the baseline
  For simple reaction time, player is asked to press space bar as soon as he sees the x appeared on the box on the screen.
  For choice based reaction times, there will be four boxes on the screen and player is asked to press the button (z, x, b and n buttons) related to the box in which the "x" symbol appeared.
Mental rotation task | At the baseline
  there will be 3 shapes on the screen with one at the top and two at the bottom. One of the shapes on the bottom is the rotated version of the one at the top. The player will be asked to find the right one, as quickly as possible. Total number of right answers will be recorded.
Kinesiophobia measurement | At the baseline
  Tampa scale of kinesiophobia (scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.) and Fear of avoidance questionnaires (he questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.) will be conducted.
Return to sport readiness | At the baseline
  ACL-RSI (Anterior Cruciate Ligament - Return to Sports after Injury: the survey consists of 12 items that are graded on a visual analogue scale from 0 points (extremely negative psychological responses) to 100 points (no negative psychological responses). The results of the survey have been found to be strongly and significantly associated with return to sport.) scoring will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Tüzün Fırat, Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosch D, Hodgson R, Peterson TL, Graf-Baumann T, Junge A, Chomiak J, Dvorak J. Assessment and evaluation of football performance. Am J Sports Med. 2000;28(5 Suppl):S29-39. doi: 10.1177/28.suppl_5.s-29. PMID 11032105
- [Background] Stoet G. PsyToolkit: a software package for programming psychological experiments using Linux. Behav Res Methods. 2010 Nov;42(4):1096-104. doi: 10.3758/BRM.42.4.1096. PMID 21139177
- [Background] Kessels RP, van Zandvoort MJ, Postma A, Kappelle LJ, de Haan EH. The Corsi Block-Tapping Task: standardization and normative data. Appl Neuropsychol. 2000;7(4):252-8. doi: 10.1207/S15324826AN0704_8. PMID 11296689
- [Background] Davis L, Appleby R, Davis P, Wetherell M, Gustafsson H. The role of coach-athlete relationship quality in team sport athletes' psychophysiological exhaustion: implications for physical and cognitive performance. J Sports Sci. 2018 Sep;36(17):1985-1992. doi: 10.1080/02640414.2018.1429176. Epub 2018 Jan 23. PMID 29359646
- See also: website from which the cognitive tests will be applied. — https://www.psytoolkit.org/